CLINICAL TRIAL: NCT05809999
Title: A Randomized Controlled Non-Inferiority Trial Comparing Neoplasia Detection During Colonoscopy Screening With and Without Non-Targeted Biopsies in Adult Colonic Inflammatory Bowel Disease
Brief Title: IBD Neoplasia Surveillance RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CTO1769
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Colonic Neoplasms; Inflammatory Bowel Diseases; Dysplasia
Keywords: Inflammatory Bowel Disease; Dysplasia; Biopsy; Colonoscopy
MeSH Terms: conditions — Colonic Neoplasms; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Participants will undergo standard colonoscopy as part of their routine IBD surveillance. During this colonoscopy targeted biopsies (biopsies of any pre-cancerous lesions observed by the doctor) and/or removal of any polyps will be undertaken.
  Interventions: Procedure: Standard colonoscopy with targeted biopsies
- Control Group (No Intervention): Participants will undergo standard colonoscopy as part of their routine IBD surveillance. During this colonoscopy both random (approximately 32 to 40) and targeted biopsies (and/or removal of any polyps) will be undertaken.

INTERVENTIONS:
Procedure: Standard colonoscopy with targeted biopsies — Participants will undergo standard colonoscopy as part of their routine IBD surveillance. During this colonoscopy targeted biopsies (biopsies of any pre-cancerous lesions observed by the doctor) and/or removal of any polyps will be undertaken.
  Arms: Experimental: Intervention Group

SUMMARY:
We will conduct a multicenter, parallel-group, non-inferiority RCT in persons with IBD undergoing colorectal neoplasia screening with high-definition white light colonoscopy, comparing a strategy of sampling visible lesions alone to a conventional strategy of sampling both visible lesions as well as normal-appearing mucosa using non-targeted biopsies. The primary outcome is the neoplasia detection rate. The required sample size to demonstrate non-inferiority is 1952 persons.

ELIGIBILITY:
Inclusion Criteria:

* Each potential participant must satisfy all of the following criteria to be enrolled in the study.

  * ≥ 18 years old
  * Historical endoscopic/histologic disease extending beyond the rectum in UC or involving ≥ 1/3 of colorectum in CD> 50% of colon present, with remaining colon meeting above minimum criteria for disease extent (beyond rectum in UC, ≥1/3 colorectum in CD)
  * cIBD ≥ 8 years duration (or at any time after diagnosis if a patient also has primary sclerosing cholangitis)
  * In symptomatic remission at time of colonoscopy

    * For CD: Harvey-Bradshaw Index < 541
    * For UC or IBDU: Partial Mayo Score ≤ 242
  * Major purpose of colonoscopy is neoplasia screening/surveillance
  * Undergoing colonoscopy with high-definition white light endoscopy

Exclusion Criteria:

* Persons who are unable to provide informed consent
* Persons with a history of colorectal cancer
* Persons with prior subtotal or total colectomy (>50% of colon removed)
* Persons undergoing repeat colonoscopy to follow-up on recently diagnosed neoplasia identified within the past year
* Persons undergoing pancolonic chromoendoscopy or pancolonic virtual chromoendoscopy
* Colon mucosa visibility deemed inadequate for surveillance after washing/suctioning (Boston Bowel Preparation Score of 0 or 1 in any segment)
* Incomplete colonoscopy (unable to reach cecum or terminal ileum [if no cecum])
* Moderate-to-severe inflammation (Mayo 2-3) involving ≥ 25% of colorectum or mild inflammation (Mayo 1) involving ≥ 50% of colorectum

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1952 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of persons with ≥ 1 neoplastic lesion detected | 4 years

SECONDARY OUTCOMES:
Mean number of neoplastic lesions per person | 4 years
Proportion of persons with ≥ 1 high grade dysplastic lesion or colorectal cancers detected | 4 years
Mean # high grade dysplastic lesions or colorectal cancers per person | 4 years
Mean # tissue samples per person | 4 years
Mean procedure time | 4 years
Rate of major adverse events within 2 weeks of procedure (as per pilot study) | 4 years
Proportion of persons referred for colectomy based on neoplastic findings | 4 years
Mean time to next recommended surveillance examination | 4 years
CRC incidence over five years following study colonoscopy (obtained through patient linkage to provincial cancer registries five years following trial completion) | 4 years

CONTACTS AND LOCATIONS:
Locations (11):
- Canada (11):
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - University of Manitoba, Health Sciences Centre, Winnipeg, Manitoba
  - Eastern Regional Health Authority, St. John's, NFLD
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec